CLINICAL TRIAL: NCT00181285
Title: Chest Wall Oscillation for Asthma and COPD Exacerbations Trial (COAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14831A
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD); Undifferentiated Asthma/COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham high frequency chest wall oscillation (Sham Comparator): Sham high frequency chest wall oscillation
  Interventions: Device: High Frequency Chest Wall Oscillator
- Active high frequency chest wall oscillation (Active Comparator): Active high frequency chest wall oscillation
  Interventions: Device: High Frequency Chest Wall Oscillator

INTERVENTIONS:
Device: High Frequency Chest Wall Oscillator — High velocity, low amplitude oscillatory airflow applied through a pneumatic vest worn over the thorax

SUMMARY:
The objective of this study was to evaluate the use of high frequency chest wall oscillation (HFCWO) early in the treatment of adults hospitalized for acute asthma or chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Acute asthma and chronic obstructive pulmonary disease (COPD) are exceedingly common, which together account for nearly 1 million hospitalizations each year in the United States alone. Beta agonists, anticholinergics, and corticosteroids delivered in aerosolized forms (via respiratory inhalers or nebulization) are recommended in the treatment of acute asthma and COPD. These medications rely on deposition into distal airspaces to suppress airway inflammation or promote bronchodilation. Unfortunately, excessive mucous production and impaired airway mucociliary clearance can lead to airway plugging, and thereby reduce the deposition of and response to aerosolized medications. These considerations highlight the need for therapies that clear airways of mucus in the acute management of asthma and COPD. High frequency chest wall oscillation (HFCWO) creates high velocity, low amplitude oscillatory airflows when applied through a pneumatic vest worn over the thorax, and is used for airway mucus clearance in patients with cystic fibrosis, bronchiectasis, and neuromuscular disorders.

This was a randomized, multi-center, double-masked phase II clinical trial of active or sham treatment initiated within 24 hours of hospital admission for acute asthma or COPD at four academic medical centers. Patients received active or sham treatment for 15 minutes three times a day for four treatments. Medical management was standardized across groups. The primary outcomes were patient adherence to therapy after four treatments (minutes used/60 minutes prescribed) and satisfaction. Secondary outcomes included change in Borg dyspnea score (≥ 1 unit indicates a clinically significant change), spontaneously expectorated sputum volume, and forced expired volume in 1 second.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Admission to the inpatient medical service
* Physician-diagnosed asthma or asthma/COPD or COPD exacerbation.
* Evidence of airflow obstruction on spirometry

Exclusion Criteria:

* More than 24 hours since admission to the inpatient medical service
* Admission to an intensive care unit
* Hospital discharge planned within the next 24 hours
* Other chronic respiratory disease (e.g., sarcoidosis, idiopathic pulmonary fibrosis)
* Chest wall abnormalities (e.g., severe kyphoscoliosis) that precludes using the vest
* Chest wall or abdominal trauma/surgery in the past 6 weeks that precludes using the vest
* Physician declines to provide consent
* Patient unable (e.g., history of cognitive impairment, unable to understand English) or declines to provide consent
* Previous participant in this study
* Corticosteroid therapy (prednisone >0 mg/d equivalent) for >1 week prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Krishnan, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Mercy Hospital and Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Mahajan AK, Diette GB, Hatipoglu U, Bilderback A, Ridge A, Harris VW, Dalapathi V, Badlani S, Lewis S, Charbeneau JT, Naureckas ET, Krishnan JA. High frequency chest wall oscillation for asthma and chronic obstructive pulmonary disease exacerbations: a randomized sham-controlled clinical trial. Respir Res. 2011 Sep 10;12(1):120. doi: 10.1186/1465-9921-12-120. PMID 21906390

RESULTS

PARTICIPANT FLOW:
Groups:
- Active High Frequency Chest Wall Oscillation: High frequency chest wall oscillation
  High Frequency Chest Wall Oscillator: High velocity, low amplitude oscillatory airflow applied through a pneumatic vest worn over the thorax
Period: Overall Study
Arm/Group | Sham High Frequency Chest Wall Oscillation | Active High Frequency Chest Wall Oscillation
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham High Frequency Chest Wall Oscillation | Active High Frequency Chest Wall Oscillation | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.4 [43.9 to 60.7] | 46.5 [38.6 to 52.8] | 48.5 [41.1 to 55.3]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender was not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Adherence to High Frequency Chest Wall Oscillation
Description: Patient adherence to therapy after four treatments.
Time Frame: After four treatments of 15 minutes each
Measure: Mean (Standard Deviation); unit: Percent of 60 minutes prescribed
Arm/Group | Sham High Frequency Chest Wall Oscillation | Active High Frequency Chest Wall Oscillation
Number analyzed (Participants) | 27 | 25
Percent of 60 minutes prescribed | 93 (18.7) | 91 (21.1)

2. Primary Outcome: Number of Participants Who Considered the Pneumatic Vest Convenient to Use
Description: The study vest was convenient to use.
Time Frame: After four treatments of 15 minutes each
Population: 1 participant in the Sham group and 1 participant in the Active group had missing data for the question regarding the convenience of the pneumatic vest, therefore these participants were not included in the number analyzed for the outcome measure data table below.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham High Frequency Chest Wall Oscillation | Active High Frequency Chest Wall Oscillation
Number analyzed (Participants) | 26 | 24
Participants | 24 | 19

ADVERSE EVENTS:
Arm/Group | Sham High Frequency Chest Wall Oscillation | Active High Frequency Chest Wall Oscillation
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No